CLINICAL TRIAL: NCT05851495
Title: Evaluation of Different Exercise Trainings Applied in Patients With Chronic Pain From Exercise Adherence, Clinical and Economic Perspectives
Brief Title: Different Exercise Trainings in Patients With Chronic Pain From Exercise Adherence, Clinical and Economic Perspectives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Irfan Kucukoglu, PhD Student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hkuirfankucukoglu001
Record Dates: First submitted 2022-12-22; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: low back pain; neck pain; exercise adherence; exercise compliance; cost effectiveness analysis; cost utility analysis; economic evaluation; icremental cost effectiveness ratio
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home-based exercise groups (No Intervention): home exercise brochures were given to the home-based exercise groups according to their diagnosis at the end of the treatment. Then, all patients were called to the hospital for control after three months and the scale prepared by us and consisting of a total of 5 (five) questions was directed to the patients and it was determined how the exercises given were performed. Five different exercises were given to patients with low back and neck pain who participated in our study. The patients were asked to do these exercises 3 times a day for 10 repetitions. Cat-camel exercises, lumbar stretching, sit-ups, bridge building and back extensor strengthening exercises were given to patients with low back pain. For patients with neck pain, neck flexion-extension, neck lateral flexion, neck rotation, shoulder capsule stretching and shoulder flexion exercises were given.
- physiotherapists-led groups (Experimental): The group involved in physiotherapists-led groups was shown the exercises in practice and under the supervision of the physiotherapist, the patients applied their exercises throughout their treatment. Then, all patients were called to the hospital for control after three months and the scale prepared by us and consisting of a total of 5 (five) questions was directed to the patients and it was determined how the exercises given were performed. Five different exercises were given to patients with low back and neck pain who participated in our study. The patients were asked to do these exercises 3 times a day for 10 repetitions. Cat-camel exercises, lumbar stretching, sit-ups, bridge building and back extensor strengthening exercises were given to patients with low back pain. For patients with neck pain, neck flexion-extension, neck lateral flexion, neck rotation, shoulder capsule stretching and shoulder flexion exercises were given.
  Interventions: Procedure: physiotherapist-led groups, home-based follow up groups
- home-based follow up groups (Experimental): Home-based follow up groups, after the exercise training was given to the patients with a physiotherapist, daily text messages (SMS) were sent to the patients and the patients were reminded to do the exercises. Then, all patients were called to the hospital for control after three months and the scale prepared by us and consisting of a total of 5 (five) questions was directed to the patients and it was determined how the exercises given were performed. Five different exercises were given to patients with low back and neck pain who participated in our study. The patients were asked to do these exercises 3 times a day for 10 repetitions. Cat-camel exercises, lumbar stretching, sit-ups, bridge building and back extensor strengthening exercises were given to patients with low back pain. For patients with neck pain, neck flexion-extension, neck lateral flexion, neck rotation, shoulder capsule stretching and shoulder flexion exercises were given.
  Interventions: Procedure: physiotherapist-led groups, home-based follow up groups

INTERVENTIONS:
Procedure: physiotherapist-led groups, home-based follow up groups — The group involved in physiotherapists-led groups was shown the exercises in practice and under the supervision of the physiotherapist, the patients applied their exercises throughout their treatment. Home-based follow up groups, after the exercise training was given to the patients with a physiotherapist, daily text messages (SMS) were sent to the patients and the patients were reminded to do the exercises
  Arms: home-based follow up groups; physiotherapists-led groups

SUMMARY:
This study was conducted with 519 patients in order to examine the clinical and cost-effectiveness of different exercise trainings in patients with chronic pain and the adherence of the patients to the exercises given. The patients were divided into 3 groups as home-based exercise groups, physiotherapist-led groups and home-based follow up groups, and traditional physical therapy was applied for a total of 10 sessions. The patients were offered exercises in the form of a brochure to the home-based exercise groups, applied to the exercise group under the guidance of a physiotherapist, and to the home-based follow up groups in a way that reminded them of the exercises by sending a daily text message (SMS) after they were given exercise training accompanied by a physiotherapist. They were told to continue their exercises after the treatment. All groups were evaluated in terms of economic, clinical, quality of life, exercise adherence, and satisfaction three times: before the treatment, after the treatment, and three months after the treatment. Cost utility analysis (QALY) and cost-effectiveness ratio (ICER) were used as part of the economic evaluation. Oswestry Disability Index (ODI) and Neck Disability Index (NDI) were used for clinical evaluation. Quality of life was assessed with the EuroQol General Quality of Life Scale (EQ-5D-5L). A scale consisting of 5 (five) questions prepared by us was used for adherence with the exercise. In the evaluation of satisfaction, individuals were asked to give a score between 0-100. All three groups were called to the hospital for control three months later, and the 5-question scale prepared by us was directed to the patients and it was determined how the given exercises were done.

DETAILED DESCRIPTION:
This study was conducted to examine the clinical and cost-effectiveness of different exercise trainings in patients with chronic pain and the adherence of the patients to the exercises given. As a result of the findings obtained, it was carried out in order to contribute to the literature, to make suggestions to the decision makers and to determine the applicability of the exercise training given by the patients. 519 patients who were admitted to the Department of Physical Medicine and Rehabilitation T.C. Ministry of Health Kilis Prof. Dr. Alaeddin Yavaşca State Hospital with a complaint of low back and neck pain were included in the study. This study was carried out at Hasan Kalyoncu University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. Patients were randomized by closed envelope randomization method as home-based exercise groups, physiotherapist-led groups, and home-based follow up groups, respectively.

The study protocol was approved by Hasan Kalyoncu University Ethical Committee (No: 2021/063, 03.05.2021). Informed consent was obtained from all of the patients.

Inclusion criteria for the study;

* 40 years and older
* Continuing low back or neck pain for 3 months or longer
* Mini mental test score more than 24 points
* Being able to speak Turkish
* Being able to be contacted via phone
* The patients participating in the study do not receive any other physiotherapy, Exclusion criteria for the study;
* Patients diagnosed with serious pathologies that may be the main cause of chronic low back pain (presence of lumbar stenosis, spondylolisthesis, fibromyalgia, etc.)
* Patients with a history of spinal surgery
* Patients for whom physiotherapy is contraindicated

Our study was planned as a prospective, randomized controlled study. The patients were pre-assessed by the physiotherapist to determine their suitability for the inclusion criteria. The first patient, whose suitability was determined, was allowed to choose his group using the closed envelope technique, and the following patients were randomized as Group-1 (home-based exercise groups), Group-2 (physiotherapist-led groups), Group-3 (home-based follow up groups).

Patients whose suitability to the inclusion criteria was evaluated by the physiotherapist were enabled to select the group with the closed envelope technique for the first one and the subsequent patients were randomized as Group-1 (home-based exercise groups), Group-2 (physiotherapist-led groups), Group-3 (home-based follow up groups) respectively. Then, home exercise brochures were given to the home-based exercise groups according to their diagnosis at the end of the treatment. The group involved in physiotherapists-led groups was shown the exercises in practice and under the supervision of the physiotherapist, the patients applied their exercises throughout their treatment. Home-based follow up groups, after the exercise training was given to the patients with a physiotherapist, daily text messages (SMS) were sent to the patients and the patients were reminded to do the exercises. Then, all three groups were called to the hospital for control after three months and the scale prepared by us and consisting of a total of 5 (five) questions was directed to the patients and it was determined how the exercises given were performed.

Demographic information of all patients participating in this study was collected through the form prepared by us.

Assessment of Exercise Adherence and Patient Satisfaction The scale consisting of a total of 5 (five) questions prepared by us three months after the treatment for exercise adherence was directed to the patients. With these questions, the patients' adherence with the exercises given to the patients was asked, the control of whether the given exercises were done correctly was as follows: "0: forgotten, 1: unable to do, 2: correct position but wrong movement, 3: correct position and movement, no respiratory control, and 4: absolutely doing". was evaluated. It was accepted that the patients who scored 3 and 4 points from the exercises remembered the exercises.

Economic Evaluation Within the scope of the economic evaluation, cost-utility and cost-effectiveness analyzes of the treatments were made. The cost-utility analysis was calculated from the perspective of the Social Security Institution (SGK) as the ratio of the total payment to the QALY (quality adjusted life years) value. For the cost-effectiveness analysis, it was calculated with the incremental cost-effectiveness ratio (ICER). In terms of the home-based follow up groups, the cost was calculated separately by adding the fees spent for home-based follow up groups purposes in addition to the SGK package fee. The Turkish version of the EQ-5D-5L scale was used to calculate the QALY value. The QALY value was calculated by evaluating the results with Germany score weights. The reason for using Germany point weights is that there is no point weights for our country and Germany point weights are used in cost effectiveness analysis studies.

Clinical Assesment Within the scope of clinical evaluation, Oswestry Disability Index was applied to patients with low back pain and Neck Disability Index was applied to patients with neck pain, and the effectiveness of the treatments were compared.

The Oswestry Disability Index is a widely used scale that measures the functional status of individuals. This scale was first described in 1980 by Fairbank et al. (122). In this scale, which consists of 10 questions in total, each question is between 0-5 points and the highest result that can be obtained from the scale is 50 points. The total score is multiplied by 2 and expressed as a percentage. The Turkish validity and reliability study of the scale, which shows that disability increases as the score obtained from the scale increases, was conducted by Yakut et al. (123).

The Neck Disability Index is a widely used scale that measures the disability level of individuals related to neck pain. This scale was defined by Vernon and Mior in 1991 (124). Neck Disability Index; It consists of 10 sections that include pain intensity, personal care, lifting, reading, headaches, concentration, work/work, driving, sleep and leisure activities. Each question consists of 6 answer options that measure the severity of pain or limitation. Scoring is done between 0-5. The highest score is 50 and the minimum score can be 0. According to the total score; 0-4: no limitation, 5-14: mild limitation, 15-24: moderate limitation, 25-34: severe limitation, 34 and above: fully restricted (124). The Turkish validity and reliability study of the scale was performed by Telci et al. (125).

Assesment of Quality of Life Quality of life was evaluated with the Turkish version of the EQ-5D-5L scale. The scale, developed by the Western European Quality of Life Research Society (EuroQoL), was introduced by the group in 2009. The scale consists of two parts, the EQ-5D descriptor system and the EQ-VAS (visual analog scale).

EQ-5D identifier system; It consists of 5 parts: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each part has 5 options: no problem, mild problem, moderate problem, serious problem and extreme problem. The patient is asked to indicate the state of health by ticking the box next to the most appropriate statement in each of the five sections. This decision results in a 1-digit number for that part. The digits of the five parts can be combined into a five-digit number describing the patient's state of health. The 5-digit number obtained from the scale is calculated using Microsoft Excel over the formulas calculated by the EuroQoL group. The answers received from these patients are placed in the program and personal values between 0 and 1 are calculated. According to this score, a value of 0 indicates death and a value of 1 indicates excellent health.

On the Visual Analog Scale (EQ-VAS), there is a vertical line with numbers up to 0-100, and the person marks the health status he/she feels for that day as 100 points at best and 0 points at worst. Thanks to this scale, it can be used as a quantitative measure of health outcomes, reflecting the patient's own decision in the form of a record of the patient's health status (126).

The validity and reliability study for the Turkish version of the EQ-5D scale and the determination of population norm values were performed by Eser et al. (127).

Exercise Protocols Five different exercises were given to patients with low back and neck pain who participated in our study. The patients were asked to do these exercises 3 times a day for 10 repetitions. Cat-camel exercises, lumbar stretching, sit-ups, bridge building and back extensor strengthening exercises were given to patients with low back pain. For patients with neck pain, neck flexion-extension, neck lateral flexion, neck rotation, shoulder capsule stretching and shoulder flexion exercises were given.

Exercises Given to Patients with Low Back Pain

1. Cat Camel Exercise: Get up on your hands and knees. Make sure your hands are at right angles to your shoulders and your knees to your hips. First, hollow your back as much as you can and lift your head (try to get your back into a C shape.) Count to 5, straighten your back and head to straighten your spine. Then lower your head, arch your back and count to 5. This movement will help your back and abdominal muscles to become flexible and compatible with each other.
2. Lumbal Stretch Exercise: Sit on a flat surface. Bend one knee and extend the other leg straight. Try to touch the toe of the straight leg with both hands. Meanwhile, your knee should not lift off the ground and your toes should not be bent towards you. Count to 10 in the lying down position and relax.
3. Sit-up Exercise: Lie on your back and bend your knees. Get help from someone or fix it somewhere so that your feet do not get off the ground. Raise your hands forward just below your shoulder blades. Keep your back on the floor and your neck straight. Count to 10 and lie on your back.
4. Bridge Building Exercise: Lie on your back with your knees bent. Tighten your abdominal muscles. Lift your hips off the ground until they're in line with your knees and shoulders. Count to 3 and lie on your back.
5. Back Extensor Strengthening Exercise: Lie face down. Extend your arms straight forward. Count backwards to 10. If you have difficulty during this movement, someone can support you by holding your feet. If there is pain, straighten a little without too much difficulty.

Exercises Given to Patients with Neck Pain

1. Neck Flexion-Extension Exercise: Without causing excessive strain, tilt your head forward so that your chin is close to your chest. After staying in this position for 10 seconds, return to your starting position and rest for 20 seconds. Then repeat the same movement with your head facing the ceiling.
2. Neck Lateral Flexion Exercise: Tilt your head so that your right ear approaches your right shoulder without causing excessive strain and without moving your shoulder. After staying in this position for 10 seconds, return to your starting position and rest for 20 seconds. Then repeat the same movement towards your left shoulder.
3. Neck Rotation Exercise: Without causing excessive strain and without moving your shoulder, turn your head to the right so that your chin is facing your right shoulder. After staying in this position for 10 seconds, return to your starting position and rest for 20 seconds. Then repeat the same movement towards your left shoulder.
4. Shoulder Capsule Stretching Exercise: Bring one arm from your shoulder level to the opposite shoulder without bending the elbow. Feel your back muscles stretch between your shoulder blades by pushing at the elbow with your other arm. Hold this position for 10 seconds, then rest for 20 seconds to relax.
5. Shoulder Fore-Back Rotation: Standing or sitting, lift both shoulders up, pull them back well and try to join them behind. At this time, feel your back muscles energize. Repeat the movement 20 times.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older
* Continuing low back or neck pain for 3 months or longer
* Mini mental test score more than 24 points
* Being able to speak Turkish
* Being able to be contacted via phone
* The patients participating in the study do not receive any other physiotherapy,

Exclusion Criteria:

* Patients diagnosed with serious pathologies that may be the main cause of chronic low back pain (presence of lumbar stenosis, spondylolisthesis, fibromyalgia, etc.)
* Patients with a history of spinal surgery
* Patients for whom physiotherapy is contraindicated

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Exercise Adherence and Patient Satisfaction | 3 months
  The scale consisting of a total of 5 (five) questions prepared by us three months after the treatment for exercise adherence was directed to the patients. With these questions, the patients' adherence with the exercises given to the patients was asked, the control of whether the given exercises were done correctly was as follows: "0: forgotten, 1: unable to do, 2: correct position but wrong movement, 3: correct position and movement, no respiratory control, and 4: absolutely doing". was evaluated. It was accepted that the patients who scored 3 and 4 points from the exercises remembered the exercises.
Economic Evaluation | 3 months
  Within the scope of the economic evaluation, cost-utility and cost-effectiveness analyzes of the treatments were made. The cost-utility analysis was calculated from the perspective of the Social Security Institution (SGK) as the ratio of the total payment to the QALY (quality adjusted life years) value. For the cost-effectiveness analysis, it was calculated with the incremental cost-effectiveness ratio (ICER). In terms of the home-based follow up groups, the cost was calculated separately by adding the fees spent for home-based follow up groups purposes in addition to the SGK package fee. The Turkish version of the EQ-5D-5L scale was used to calculate the QALY value. The QALY value was calculated by evaluating the results with Germany score weights. The reason for using Germany point weights is that there is no point weights for our country and Germany point weights are used in cost effectiveness analysis studies.
Oswestry Disability Index | 3 months
  The Oswestry Disability Index is a widely used scale that measures the functional status of individuals. This scale was first described in 1980 by Fairbank et al. (122). In this scale, which consists of 10 questions in total, each question is between 0-5 points and the highest result that can be obtained from the scale is 50 points. The total score is multiplied by 2 and expressed as a percentage. The Turkish validity and reliability study of the scale, which shows that disability increases as the score obtained from the scale increases, was conducted by Yakut et al. (123).
Neck Disability Index | 3 months
  The Neck Disability Index is a widely used scale that measures the disability level of individuals related to neck pain. This scale was defined by Vernon and Mior in 1991 (124). Neck Disability Index; It consists of 10 sections that include pain intensity, personal care, lifting, reading, headaches, concentration, work/work, driving, sleep and leisure activities. Each question consists of 6 answer options that measure the severity of pain or limitation. Scoring is done between 0-5. The highest score is 50 and the minimum score can be 0. According to the total score; 0-4: no limitation, 5-14: mild limitation, 15-24: moderate limitation, 25-34: severe limitation, 34 and above: fully restricted (124). The Turkish validity and reliability study of the scale was performed by Telci et al. (125).
Assesment of Quality of Life | 3 months
  EQ-5D identifier system; It consists of 5 parts: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each part has 5 options: no problem, mild problem, moderate problem, serious problem and extreme problem. The patient is asked to indicate the state of health by ticking the box next to the most appropriate statement in each of the five sections. This decision results in a 1-digit number for that part. The digits of the five parts can be combined into a five-digit number describing the patient's state of health. The 5-digit number obtained from the scale is calculated using Microsoft Excel over the formulas calculated by the EuroQoL group. The answers received from these patients are placed in the program and personal values between 0 and 1 are calculated. According to this score, a value of 0 indicates death and a value of 1 indicates excellent health.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Yes